CLINICAL TRIAL: NCT03057782
Title: Innovative Approaches to Assessment of Pain Control and Sedation in the NICU
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Laura Cornelissen PhD, PhD, Boston Children's Hospital
Other Study IDs: IRB-P00022180
Record Dates: First submitted 2016-11-28; First posted 2017-02-20 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Pain, Postoperative
Keywords: Pain; Sedation; Surgery
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group A: 1. Plan for major surgery anticipated to cause pain and agitation (i.e. esophageal atresia treatment);
  2. Patients who are anticipated to receive prolonged post-surgical neuromuscular blockade (NMB)
  The following devices will be used in this Group: Waveguard (TM) EEG cap; Micro Movement Sensor; Pico Movement Sensor; QS Piezostimulator; tactileTM sensory evaluator. These subjects will also receive EMG monitoring. Subjects in this group will also have video recordings that may be used for novel analysis such as subdermal blood flow or micro-movement.
  Interventions: Device: Waveguard (TM) EEG cap; Device: Micro Movement Sensor; Device: Pico Movement Sensor; Device: QS Piezostimulator; Device: tactileTM sensory evaluator
- Group B: 1. Plan for major surgery anticipated to cause pain and agitation (i.e. bowel surgery);
  2. Patients who are not anticipated to receive acute post-surgical NMB
  The following devices will be used in this Group: Waveguard (TM) EEG cap; Micro Movement Sensor; Pico Movement Sensor; QS Piezostimulator; tactileTM sensory evaluator. Subjects in this group will also have video recordings that may be used for novel analysis such as sub-dermal blood flow or micro-movement.
  Interventions: Device: Waveguard (TM) EEG cap; Device: Micro Movement Sensor; Device: Pico Movement Sensor; Device: QS Piezostimulator; Device: tactileTM sensory evaluator
- Group C: Plan for minor surgery anticipated to cause pain and agitation (i.e. hernia repair)
  The following devices will be used in this Group: Waveguard (TM) EEG cap; Micro Movement Sensor; Pico Movement Sensor; QS Piezostimulator; tactileTM sensory evaluator. Subjects in this group will also have video recordings that may be used for novel analysis such as sub-dermal blood flow or micro-movement.
  Interventions: Device: Waveguard (TM) EEG cap; Device: Micro Movement Sensor; Device: Pico Movement Sensor; Device: QS Piezostimulator; Device: tactileTM sensory evaluator
- Group D: No plan for surgery
  The following devices will be used in this Group: Waveguard (TM) EEG cap; Micro Movement Sensor; Pico Movement Sensor; QS Piezostimulator; tactileTM sensory evaluator. Subjects in this group will also have video recordings that may be used for novel analysis such as sub-dermal blood flow or micro-movement.
  Interventions: Device: Waveguard (TM) EEG cap; Device: Micro Movement Sensor; Device: Pico Movement Sensor; Device: QS Piezostimulator; Device: tactileTM sensory evaluator

INTERVENTIONS:
Device: Waveguard (TM) EEG cap — The device is an EEG cap - a non-invasive EEG positioning system used to quickly place a large number of surface electrodes in a quick and consistent manner on the head. The device will measure electrophysiological signals from the scalp at the time points in the study listed in the protocol.
Device: Micro Movement Sensor — This device is not FDA approved. This device is in clinical use for all age groups and used for research purposes by neurologists, physiologists and anesthesiologists. In this study, the device is used to monitor breathing and movement in children; the device is not used for validation purposes.
Device: Pico Movement Sensor — This device is not FDA approved. This device is in clinical use for all age groups and used for research purposes by neurologists, physiologists and anesthesiologists. In this study, the device is used to monitor respiration rate and gross body movement in children. The device will not be used for validation purposes.
Device: QS Piezostimulator — This device is not FDA approved. This device is used for research purposes by neurologists and physiologists. It is a mechanical tactile stimulator for use in functional imaging experiments like MEG, fMRI or EEG. The stimulation is realized by using several different pin matrices. In this study, the device is used to stimulate the children's extremities in order to elicit somatosensory evoked responses.
Device: tactileTM sensory evaluator — This device is not FDA approved. This device is used for clinical and research purposes by neurologists and physiologists. It is used to stimulate the children's extremities in order to elicit somatosensory evoked responses.

SUMMARY:
It is difficult to assess pain and agitation in the NICU population because for a multitude of reasons including the pre-verbal nature of the patient population, the atypical pain response of premature infants, and the use of muscle relaxing medications that exclude motor response in pain assessments. Current assessment tools are based on physical exam and vital signs. The investigators propose to study the role of EEG and palmar conductance (PD) as additional tools in the assessment of pain and agitation

DETAILED DESCRIPTION:
This is a prospective, non-interventional study designed to assess noxious-specific neurophysiologic responses and clinical signs following procedural pain in infants requiring hospitalization in the neonatal intensive care unit (NICU) following elective surgery.

The main goal of the study is to develop a method that reliably quantifies the level of pain induced from clinically-required noxious procedures to infants hospitalized in the NICU. This method will use measures of neurophysiological, autonomic, and behavioral responses to non-noxious and clinically-required noxious stimuli in order to guide the pharmacological treatment of NICU patients with analgesic agents, sedatives and/or muscle relaxants.

The investigators hypothesize that resting state activity and physiological responses to noxious and non-noxious stimuli provide a more reliable assessment of the level of pain of infants hospitalized in the NICU compared to behavioral-based pain scores.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be admitted to the NICU, and having a post-menstrual age of >28 weeks. Participants will be divided into four groups according to the following criteria:

Group A

* Plan for major surgery anticipated to cause pain and agitation (i.e. esophageal atresia treatment);
* Patients who are anticipated to receive prolonged post-surgical neuromuscular blockade

Group B

* Plan for major surgery anticipated to cause pain and agitation (i.e. bowel surgery);
* Patients who are not anticipated to receive acute post-surgical neuromuscular blockade

Group C Plan for minor surgery anticipated to cause pain and agitation (i.e. hernia repair);

Group D No plan for surgery

Exclusion Criteria:

* Confirmed or suspected clinical seizures
* Metabolic abnormalities or inborn error of metabolism
* Skin abrasions or wounds located at the site of research sensor placement i.e. scalp, which interfere with the application of electrodes

Ages: 1 Hour to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a prospective, non-interventional study designed to assess neurophysiologic responses and clinical signs to noxious and non-noxious stimuli following procedural pain in infants requiring NICU care following elective surgery. Simultaneous measures of neurophysiological, autonomic and behavioral responses to non-noxious and clinically-required noxious stimuli will be collected from patients in the NICU.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Noxious Stimuli Results | Up to 1 year
  To assess pain-specific brain activity and autonomic responses post surgery in response to an acute noxious procedure in newborn infants admitted to the NICU. This outcome will be correlated with current behavioral and physiological based pain assessment tools as follows:
  Procedural-specific brain activity in infants with varying conditions with pre or post-operative pain. EEG: amplitude of noxious-event related potential evoked by a time-locked noxious stimulus. Pain-specific electro-dermal activity (EDA), electromyography (EMG) and subdermal skin flow; Pain-evoked behavioral measures including: Body movement; Eye squeeze, brow bulge and nasolabial furrow duration. Pain-evoked physiological measures including: Respiration rate; Heart rate; Blood pressure; Oxygen saturation; Observational pain scores (PIPP); EMG activity.

SECONDARY OUTCOMES:
Resting State Results | Up to 1 year
  Characterize resting state activity in post-operative or control subjects as follows:
  Baseline brain (EEG) activity (power spectra of baseline EEG signal) in post operative or control subjects. Baseline EDA, EMG and subdermal skin flow; Baseline behavioral measures including: Presence of body movement, eye squeeze, brow bulge and nasolabial furrow. Baseline physiological measures including: Respiration rate; Heart rate; Blood pressure; Oxygen saturation; Observational pain scores (PIPP).
  The relationship with resting brain activity, electrodermal activity, behavior, physiological, and observational pain scores will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Cornelissen, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No